CLINICAL TRIAL: NCT02107950
Title: A Randomized, Open-label, Parallel Group, Multi-center Phase II Clinical Trial DCVAC/OvCa Added to Standard Chemotherapy in Women With Relapsed Platinum Sensitive Epithelial Ovarian Carcinoma
Brief Title: Phase II Study DCVAC/OvCa Plus Carboplatin Gemcitabine Relapsed Platinum (Pt)-Sensitive Epithelial Ovarian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOV02; 2013-001323-38 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2016-01

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer (OvCa); Ovarian Epithelial Cancer
Keywords: Ovarian; Platinum Sensitive; Epithelial
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy; Carboplatin; Gemcitabine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCVAC/OvCa in parallel with chemotherapy (Experimental): Combination therapy with DCVAC/OvCa and Standard of Care
  Interventions: Biological: DCVAC/OvCa in parallel with chemotherapy
- Standard of Care (Active Comparator): Standard of Care carboplatin and gemcitabine
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Biological: DCVAC/OvCa in parallel with chemotherapy — DCVAC/OvCa is the experimental therapy added on to Carboplatin and Gemcitabine
  Other Names: DCVAC/OvCa; carboplatin and gemcitabine
  Arms: DCVAC/OvCa in parallel with chemotherapy
Drug: Standard of Care — Carboplatin and Gemcitabine is Standard of Care First Line Chemotherapy
  Other Names: Carboplatin and Gemcitabine
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine whether DCVAC/OvCa added to chemotherapy (carboplatin and gemcitabine as second line chemotherapy) may result in prolongation of progression free survival (PFS).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether DCVAC/OvCa added to Standard of Care chemotherapy (carboplatin and gemcitabine as second line chemotherapy) may result in prolongation of progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years old and older
* Patients with histologically confirmed, International Federation of Gynecology and Obstetrics (FIGO) stage III or IV epithelial ovarian, primary peritoneal or fallopian tube carcinoma (serous, endometrioid or mucinous), who had complete remission after first line platinum (Pt)-based chemotherapy and are selected to receive second line Standard of Care chemotherapy
* Radiologically confirmed relapse after >6 months of remission (Platinum-sensitive patients), found up to 4 weeks prior study entry.
* The patient must have at least one measureable target lesion as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria to be eligible for enrolment in the study

Exclusion Criteria:

* FIGO I,II epithelial ovarian cancer
* FIGO III, IV clear cells epithelial ovarian cancer
* Non-epithelial ovarian cancer
* Borderline tumors (tumors of low malignant potential)
* Prior or current systemic anti-cancer therapy for ovarian cancer [for example chemotherapy, monoclonal antibody therapy , tyrosine kinase inhibitor therapy, vascular endothelial growth factor (VEGF) therapy or hormonal therapy] except first line Platinum-based chemotherapy (with or without bevacizumab)
* Previous radiotherapy to the abdomen and pelvis
* Malignancy other than epithelial ovarian cancer, except those that have been in clinical remission (CR) for a minimum of 3 years, and except carcinoma in-situ of the cervix or non-melanoma skin carcinomas

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Determine median progression free survival | 72 Week

SECONDARY OUTCOMES:
Overall survival (all causes) | 56, 64, 72 weeks
Objective Response Rate | 8, 16, 24, 32, 40, 48, 56. 64. 72 weeks
Biological Progression Free Interval | 6, 12, 18, 24, 36, 42, 48, 56, 64, 72 weeks
Immunological Response | 24, 48, 72 weeks
Frequency of adverse events | 8, 16, 24, 32, 40, 48, 56. 64. 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ales Horacek, Study Director — Accord Research
Locations (14):
- Czechia (7):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Nový Jičín
  - Olomouc
  - Ostrava
  - Prague
- Germany (3):
  - Cologne
  - Dresden
  - Erlangen
- Poland (4):
  - Bialystok
  - Krakow
  - Lublin
  - Poznan

IPD SHARING:
Plan to Share IPD: Yes
will be posted to EMA website
Supporting Information: Study Protocol, CSR
Time Frame: estimate end of 2018

REFERENCES:
- [Derived] Cibula D, Rob L, Mallmann P, Knapp P, Klat J, Chovanec J, Minar L, Melichar B, Hein A, Kieszko D, Pluta M, Spacek J, Bartos P, Wimberger P, Madry R, Markowska J, Streb J, Valha P, Hassan HIB, Pecen L, Galluzzi L, Fucikova J, Hrnciarova T, Hraska M, Bartunkova J, Spisek R. Dendritic cell-based immunotherapy (DCVAC/OvCa) combined with second-line chemotherapy in platinum-sensitive ovarian cancer (SOV02): A randomized, open-label, phase 2 trial. Gynecol Oncol. 2021 Sep;162(3):652-660. doi: 10.1016/j.ygyno.2021.07.003. Epub 2021 Jul 20. PMID 34294416